CLINICAL TRIAL: NCT07282665
Title: A PHASE 3, PLACEBO-CONTROLLED, DOUBLE-BLINDED, RANDOMIZED STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF A CLOSTRIDIOIDES DIFFICILE VACCINE IN ADULTS 65 YEARS OF AGE AND OLDER
Brief Title: A Study to Learn About a Clostridioides Difficile Vaccine in People 65 Years of Age and Older
Acronym: BEETHOVEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4771002
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Clostridioides Difficile Associated Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- C.difficile vaccine (Experimental): Novel vaccine formulation
  Interventions: Biological: C.difficile vaccine
- Saline Placebo (Other)
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Biological: C.difficile vaccine — C.difficile vaccine given as an intramuscular injection
  Arms: C.difficile vaccine
Other: Saline Placebo — 0.9% sodium chloride solution given as a intramuscular injection
  Arms: Saline Placebo

SUMMARY:
The purpose of the study is to learn about how effective, safe, and tolerable the Clostridioides difficile (C. difficile) vaccine is in decreasing the number of C. difficile infections (pCDI) in adults 65 years of age or older.

The participants will receive either the C. difficile vaccine or placebo (saline). A placebo does not contain any active ingredients. The vaccines will be given as a shot into the upper arm muscle.

This study looks at the number of diarrhea (loose stools) events related to a C. difficile infection, so the length of the study can change. If these events happen quickly, the study may finish sooner; if they happen slowly, it could take longer. Sometimes, the study might stop early if the vaccine clearly works or clearly doesn't. Participants will stay in the study until enough events have occurred to answer the main question. On average, each person is expected to take part for up to about three and a half years.

During this time, participants will have 3 planned clinical visits and 3 planned phone visits. After these visits, more scheduled clinic visits will happen every year until the end of study.

Besides the scheduled study visits, if at any time during the study a participant has 3 or more loose stools in 24 hours, they will be asked to save the next one (the fourth or later) and contact the study site. The study site will check to see if it could be a C. difficile infection. This check may happen at the clinic or through a phone or video call.

ELIGIBILITY:
Who Can Join the Study (Inclusion Criteria):

• People with recent or future planned contact with healthcare systems or who have recently received antibiotics.

Who Cannot Join the Study (Exclusion Criteria):

* Anyone who has had CDI before.
* Anyone who has had surgery to remove part of their small or large intestine.
* Anyone who often has diarrhea (meaning three or more loose stools in a day, more than once a month).
* Anyone who has already received a vaccine or special antibody treatment for C. difficile.
* Anyone who has had a serious allergic reaction to a vaccine or to any part of the study vaccines.
* Anyone who might not respond well to the vaccine because their immune system is weak (either from a disease or from treatment).
* Anyone with cancer that has spread, kidney failure, or another serious health problem.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32000 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2029-06-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants reporting local reactions | For 7 days after each vaccination
  Injection site pain, redness, and swelling as self-reported in electronic diaries
The percentage of participants reporting systemic events | For 7 days after each vaccination
  Fever, vomiting, fatigue, headache, muscle pain, and joint pain as self-reported in electronic diaries
Percentage of participants reporting adverse events | From each vaccination through 1 month after each vaccination
  As elicited by investigator site staff
Percentage of participants reporting serious adverse events | From Vaccination 1 (Day 1) through 12 months after Vaccination 2 (last dose) (18 months)
  As elicited by investigator site staff
The incidence of the first episode of medically attended and clinically meaningful primary Clostridioides difficile infection (CDI) | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of medically attended and clinically meaningful primary CDI incidence per 1000 person- years of follow- up
The incidence of the first episode of medically attended primary CDI | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of medically attended primary CDI incidence per 1000 person- years of follow- up
The incidence of the first episode of clinically meaningful primary CDI | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of clinically meaningful primary CDI incidence per 1000 person- years of follow- up

SECONDARY OUTCOMES:
The incidence of antibiotic use in the treatment of a first episode of the primary CDI | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of primary CDI with antibiotic use incidence per 1000 person- years of follow- up
The incidence of severe primary CDI as defined by Infectious Diseases Society of America (IDSA)/ Society for Healthcare Epidemiology of America (SHEA) | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of severe or fulminant primary CDI incidence per 1000 person- years of follow- up
The incidence of a first episode of primary CDI (any severity) | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  First episode of primary CDI incidence per 1000 person- years of follow- up
The incidence of all CDI (primary and recurrent) | from 14 days after Vaccination 2 to the end of the surveillance period (up to approximately 3.5 years)
  Time to all C.difficile infection cases

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (83):
- United States (68):
  - North Alabama Research Center, Athens, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Epic Medical Research-Sun City, Sun City, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Velocity Clinical Research, San Bernardino, San Bernardino, California
  - Carbon Health - San Mateo - Hillsdale Mall, San Mateo, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - GW Vaccine Research Unit, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - M3 Wake Research - Lake City, Lake City, Florida
  - South Florida Research Organization, Medley, Florida
  - Care Research Inc, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - DM Clinical Research - Chicago, Melrose Park, Illinois
  - Accellacare - McFarland, Ames, Iowa
  - McFarland Clinic, PC, Ames, Iowa
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - AMR Clinical, Newton, Kansas
  - Revive Research Institute, Inc., Southfield, Michigan
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Renown Center for Advanced Medicine, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - University Health, Reno, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Upstate Global Health Institute, East Syracuse, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Cary, Cary, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Walker Family Care, Little River, South Carolina
  - Trial Management Associates, LLC, Myrtle Beach, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Family Health Watch - KeyPoint Clinical Research, Dallas, Texas
  - KeyPoint Clinical Research, Dallas, Texas
  - Cedar Health Research - Euless, Euless, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - Mercury Clinical Research - Santa Clara Family Clinic, Houston, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
  - University of Washington - Harborview Medical Center, Seattle, Washington
- Argentina (2):
  - Equipo Ciencia, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Sagrado Corazón, Buenos Aires
- United Kingdom (13):
  - Newquay Health Centre, Newquay, Cornwall
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Knowle House Surgery, Plymouth, Devon
  - Brunel Medical Practice (St Marychurch), Torquay, Devon
  - Panthera Biopartners - Preston, Preston, England
  - Synexus Scotland Clinical Research Centre, Glasgow, Glasgow CITY
  - Panthera Biopartners - Manchester, Rochdale, Manchester
  - Panthera Clinic - York, York, North Yorkshire
  - Lakeside Surgery, Corby, Northamptonshire
  - Panthera Biopartners - Glasgow, Glasgow, Scotland
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Synexus Manchester Clinical Research Centre, Manchester
  - Panthera Biopartners - Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4771002